CLINICAL TRIAL: NCT04307849
Title: Engaging Providers, Community Members, and Young Women to Adapt and Pilot a Youth-friendly Sexual and Reproductive Health Package in Low-income Communities in India
Brief Title: Youth-friendly Sexual and Reproductive Healthcare Pilot in Mumbai, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-00240; 1K01TW011480-01 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-03-13 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Reproductive Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescent Health Club (Experimental): A systematic approach for the adaptation of sexual health/HIV-related evidence-based interventions
  Interventions: Behavioral: Adolescent Health Club
- Wait-list Control (Placebo Comparator)
  Interventions: Behavioral: Adolescent Health Club; Other: Wait-list Control

INTERVENTIONS:
Behavioral: Adolescent Health Club — Sexual health/HIV-related evidence-based interventions
Other: Wait-list Control — The wait-listed group will begin the intervention after the intervention group
  Arms: Wait-list Control

SUMMARY:
This study will systematically adapt, pilot test, and evaluate an integrated community/facility intervention to improve the uptake of adolescent-friendly services for married and unmarried adolescent girls and young women (AGYW; ages 15-25) in a low-income area with a population of approximately 700,000 in Mumbai, India

DETAILED DESCRIPTION:
Aim 1: Adapt the health club curriculum and provider/staff sensitization training using Assessment, Decision, Administration, Production, discussion with Topical experts, Integration, Training, and Testing (ADAPT-ITT) Formative mixed methods data will be collected from stakeholders to assess the landscape of adolescent-friendly care and gaps to adapt the intervention. Intervention sessions will be presented to groups of stakeholders to elicit feedback on adaptations.

The formative research entails a mixed methods assessment of the adolescent sexual reproductive health landscape in the study area, and adaptation of the intervention components through interactive sessions, consistent with ADAPT-ITT.

ADAPT-ITT Assessment Phase

Key informant interviews (KIIs) - Qualitative key informant interviews (N=35) will be conducted with both public and private community-based health providers, NGO workers, community health workers (CHWs), and parents of young women. Interviews will also be conducted with government officials at the community and M Ward levels (wards are the smallest administrative unit of governmental ministries). These interviews will focus on qualitative mapping of adolescent health and treatment-seeking pathways and providers in the study area, and factors in the family, community, and elsewhere that influence adolescent girls' and young women's health. The KIIs will also provide insight into aspects of the intervention and evaluation tools requiring modification. KIIs will also be invited to join a community advisory board (CAB) for the duration of the project. This CAB will provide a forum for AGYW to present their learnings from the adolescent club, and serve as a resource should community members have questions or concerns about the intervention.

In-depth interviews with adolescent girls and young women (IDIs) - Qualitative in-depth interviews will be conducted with 20 AGYW (aged 15-25 years old) to understand their experiences with healthcare in the study area, treatment-seeking patterns, and factors in the family, community and elsewhere that influence their health. Young women will also be asked to comment on the proposed intervention's feasibility and acceptability, and provide input on aspects of the intervention and evaluation tools that need modification. Roughly equal numbers of married and unmarried young women will be recruited for participation. Young women will be recruited with assistance from NGO programs, CHWs, and referrals from other participants.

Survey with AGYW on care-seeking patterns and perceptions of healthcare quality and quantitative analysis - A random sample of AGYW seeking care at a set of public (N=3) and private (N=3) healthcare facilities in the study area will be selected and asked to participate in a brief, 20-30 minute survey using validated measures to discuss their patterns of healthcare-seeking (where they go for different problems, and what influences those choices), and their perceptions and experiences with adolescent healthcare. For unmarried participants under the age of 18, consent will be obtained from both a parent and the young woman. The investigators involved in this study have experience obtaining consent from parents, and do not anticipate challenges obtaining consent. About 20-25 AGYW will be surveyed from each facility, with a total N=100-150. Survey data will be entered into R, and bivariate and multivariate analyses will be conducted to understand factors associated with AGYW treatment-seeking that may need to be addressed in the health clubs. Analyses will also explore quality of care to identify elements that may need to be incorporated into the provider sensitization. This survey will the investigators to apply skills gained in Training Aim 1.

Theater testing with key stakeholders for intervention adaptations - Theater testing meetings will be held in which intervention sessions are presented and, in some cases, acted out to the group. Audience members' responses and post-meeting critiques of the material will be recorded and analyzed (see below). During the meetings, both general feedback, as well as whether adolescent health club sessions need to be conducted separately with different age groups or based on marital status (married adolescents, regardless of age could have different needs than unmarried adolescents) will be evaluated. Separate meetings will be held with the following stakeholder groups to present the intervention modules and elicit feedback on revisions or adaptations: 1) AGYW; 2) community members/KIIs; and 3) healthcare providers, CHVs, and NGO staff. Additional meetings may be conducted after modifications are made to ensure agreement

Qualitative data analysis and finalization of intervention modules - Interviews and group discussions will be transcribed and translated (as needed, some KII materials will already be in English) and coded with the qualitative data analysis software, Atlas.ti. Using a framework approach with codes based on key implementation and conceptual model factors of interest, data will be coded and analyzed to identify elements of the intervention needing revision, with additional codes added as novel topics/issues arise.Coding will be conducted by myself and a research assistant, consulting with Dr. Maitra as needed. Using the formative data and the expertise of my mentors, the intervention modules will be adapted to the context, while making sure the key evidence-based elements are not lost. As needed, additional in-depth coding of the formative qualitative data can be conducted once rapid analysis for intervention adaptation has been completed. Once the modules have been finalized, the intervention facilitators will be trained, and the intervention implemented.

Aim 2: Implement a pilot of the intervention and assess implementation outcomes.

The provider and staff component will consist of two groups to facilitate participation and accommodate provider/staff schedules. Four separate groups of AGYW will participate in the adolescent health club component, using a wait-list control group design. Separate groups are needed due to the group nature of the intervention activities which limits the number of people who can participate at one time. Intervention participants will be surveyed pre- and post-intervention to examine acceptability, feasibility, and uptake. Qualitative process data will also be collected and analyzed.

Aim 3: Assess a pilot set of health outcomes for future research. Quantitative pre- and post-tests will also assess pilot effectiveness health and behavioral outcomes.

Intervention (the "Testing" phase of ADAPT-ITT: Research Aims 2 and 3)

The ADAPT-ITT Model - The ADAPT-ITT model was developed by Wingood and DiClemente as a systematic approach for the adaptation of sexual health/HIV-related evidence-based interventions.41 The ADAPT-ITT acronym stands for each of the eight phases of the model (although not all applications of the model use all phases): assessment, decision, administration, production, discussion with topical experts, integration, training, and testing. The assessment phase involves conducting needs assessments with the target population. The decision phase (which for some studies, such as the one proposed here, happens before the assessment) occurs when one chooses the evidence-based intervention(s) to be adapted. Administration involves the use of theater tests or interactive presentations with key stakeholders to determine what adaptations are needed and to ensure the intervention will be designed with end-users in mind. The revised/adapted draft of the intervention is finalized in the production and integration phases with the guidance of topical experts and information from the theater tests. Once the research team is trained in intervention delivery, the intervention can be pilot tested and results analyzed. The model explicitly includes the target population/patients/end-users and other key stakeholders in the process of intervention adaptation, enabling a participatory approach to implementation. Not all frameworks or models of implementation allow for this engagement, which is why the ADAPT-ITT approach was chosen. The ADAPT-ITT model has been used to adapt interventions for sexual and reproductive health substance use,mental and behavioral health, and chronic health issues in both international and domestic settings.

Neither providers/staff or clinics can be randomized, as only a subset of the clinics/providers in the study area see enough AGYW to meet inclusion criteria, and some providers/staff who participate will work in the same clinics. Providers/staff will complete brief pre- and post-training surveys; however, the primary measures of their intervention will be derived from the AGYW's outcomes.

For the adolescent health club component, the pilot study employs a waitlisted control group design. In this modified version of the stepped wedge design, all groups receive the intervention, and participants serve as their own controls. This design utilizes a smaller sample size of AGYW and fewer facilitators, making it more feasible for a K award, while still enabling all participants to participate in the intervention. The waitlisted control design also avoids some of the challenges associated with carryover effect that can occur in other crossover designs, as participants move unidirectionally from control to intervention. The adolescent health club curriculum (which takes approximately 2.5 months to complete) will be sequentially administered to four groups, each with a waitlisted control group. Individuals can be compared to themselves, and the other groups. Sequentially administering the intervention will be more feasible than administering the intervention simultaneously to separate neighborhood clusters, limiting the number of facilitators needed.

Provider Sensitization Component and Evaluation - Providers and clinic staff at the public UHC and health posts, as well as from private clinics known to provide care for adolescents will be screened to determine if they meet eligibility criteria, and if they do, then they will be invited to participate in the sensitization workshop. There will be two workshop groups with 20 participants each. All participants will complete pre/post intervention surveys, primarily focused on feasibility and acceptability of the intervention, using previously validated measures. After each session, the facilitator will complete a log to code activities as implemented fully, implemented partially or modified significantly and describe any changes. The log will also include a section to document any unusual events associated with any of the sessions, and the effect of these events on implementation, acceptability, or feasibility. Every other session will be observed and documented in fieldnotes that will be analyzed to contribute to process evaluation (see analysis details below). The log and observations will enable a qualitative assessment of intervention fidelity. A subset will be selected for exit interviews to contextualize the quantitative measures, and learn about participants' perspectives on feasibility and acceptability.

Adolescent Health Club Component and Evaluation - Households with AGYW ages 15 to 25 will be identified by community health workers from randomly selected block sectors of the study area. Clubs will be conducted in separate neighborhood sectors, to limit contamination. Conducting club meetings near to the lanes adolescent girls live in will make it easier for attendance. To further assess and address potential contamination, individuals will be asked to verify the adolescent health club they attended in the post-intervention survey, whether they attended an additional health club outside the intervention (such as, in school). If any contamination is evident based on this question, it will be modeled in the analysis. AGYW and their mothers (if unmarried and under the age of 18) will be approached by a member of the research team and the adolescent health club intervention will be explained. If consent is obtained, the AGYW will be enrolled, and randomized to either participate or join the wait-list. AGYW will complete the pre-intervention evaluation instrument upon enrollment. In addition to the activities in the "It's All One" Curriculum spread over eight modules, providers from the sensitization component will attend one meeting to discuss services available in the adolescent-friendly clinics, and hear young women's previous experiences accessing care. Similar to the process for the provider sensitization component, the facilitator will complete a log after each session to code activities as implemented fully, implemented partially or modified significantly and describe any changes. The log will also include a section to document any unusual events associated with any of the sessions, and the effect of these events on implementation, acceptability, or feasibility. Every other session will be observed and documented in fieldnotes that will be analyzed to contribute to process evaluation (see analysis details below). As with the provider component, the log and fieldnotes will enable a qualitative assessment of intervention fidelity. When young women complete the curriculum, they will also complete the post-intervention evaluation instrument. A sub-sample of young women (N=15) will be asked to participate in a focus group discussion to reflect on the club's impact and acceptability. Domains measured by previously validated instruments to be covered in the pre- and post-intervention surveys. There are relatively few validated quantitative measures of implementation outcomes, and none in Hindi, thus the measure chosen will have to be translated and back-translated to ensure comprehension.

ELIGIBILITY:
Inclusion Criteria:

* AGYW between the ages of 15-25 years old
* Provide consent or assent,
* Living in the study area for one year or more,
* If unmarried and under the age of 18, have parental consent to participate. Married AGYW and/or those age 18 or over will be recruited if they meet inclusion criteria and provide informed consent.

Exclusion Criteria:

* AGYW who are unable to give consent due to psychological or mental limitations,
* If unmarried and under the age of 18 do not have parental consent to participate.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Brault, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- Apnalaya, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wingood GM, DiClemente RJ. The ADAPT-ITT model: a novel method of adapting evidence-based HIV Interventions. J Acquir Immune Defic Syndr. 2008 Mar 1;47 Suppl 1:S40-6. doi: 10.1097/QAI.0b013e3181605df1. PMID 18301133
- [Background] Hunsley J. Development of the treatment acceptability questionnaire. Journal of Psychopathology and Behavioral Assessment. 1992;14(1):55-64.
- [Background] Cleland J, Ingham R, Stone N. Asking young people about sexual and reproductive behaviours: Illustrative Core Instruments. World Health Organization, 2001.
- [Background] Bhatla N, Achyut P, Ghosh S, Gautam A, Verma R. Safe Cities Free From Violence Against Women and Girls: Baseline Finding from the
- [Background] Achyut P, Bhatia N, Singh A, Verma R, Khandekar S, Pallav P, et al. Building support for gender equality among young adolescents in school: findings from Mumbai India. 2011.
- [Background] Brault MA, Schensul SL, Bankar S. The role of pre-marital agency in delaying marriage and reproductive decision-making in urban India. In: Erausquin MWaJT, editor. Global Perspectives on Women's Reproductive and Sexual Health Across the Lifespan: Springer Press Publishers; 2017.
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Lewis CC, Fischer S, Weiner BJ, Stanick C, Kim M, Martinez RG. Outcomes for implementation science: an enhanced systematic review of instruments using evidence-based rating criteria. Implement Sci. 2015 Nov 4;10:155. doi: 10.1186/s13012-015-0342-x. PMID 26537706

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that parents of participants were not enrolled in the study.
Groups:
- Group A: Participants in Group A receive the intervention during Intervention Period 1 and do not have wait list control data collected.
- Group B: Participants in Group B have wait list control data collected during Intervention Period 1, and receive the intervention during Intervention Period 2.
- Group C: Participants in Group C have wait list control data collected during Intervention Period 2, and receive the intervention during Intervention Period 3.
- Group D: Participants in Group D have wait list control data collected during Intervention Period 3 and receive the intervention during Intervention Period 4.
- Physician Workshop Participants: Physicians who participate in the facility-based intervention
- Community Health Volunteers (CHV) Workshop Participants: CHVs who participate in the intervention sessions.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Physician Workshop Participants | Community Health Volunteers (CHV) Workshop Participants
Started | 25 | 25 | 25 | 25 | 41 | 20
# Participants Started Intervention Period 1: | 25 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 0 | 0 | 0
# Participants Completed Intervention Period 1: | 23 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 0 | 0 | 0
# Participants Started Intervention Period 2: | 0 | 25 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 23 | 20
# Participants Completed Intervention Period 2: | 0 | 23 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 21 | 19
# Participants Started Intervention Period 3: | 0 | 0 | 25 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 0
# Participants Completed Intervention Period 3: | 0 | 0 | 19 (Receive intervention) | 25 (Wait-list control data collected) | 0 | 0
# Participants Started Intervention Period 4: | 0 | 0 | 0 | 25 (Receive intervention) | 18 | 0
# Participants Completed Intervention Period 4: | 0 | 0 | 0 | 22 (Receive intervention) | 16 | 0
Completed | 23 | 23 | 19 | 22 | 37 | 19
Not Completed | 2 | 2 | 6 | 3 | 4 | 1
Not completed — Took a paid position and/or work schedule no longer allowed participation | 2 | 2 | 1 | 2 | 4 | 1
Not completed — Travelled out of Mumbai to natal place/village | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Family member did not want them to continue | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Medical reason (gave birth, became ill) | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Note that the data presented represents all available baseline characteristic data. No baseline data were collected from CHV workshop participants and thus are not presented here.
Groups:
- Physician Workshop Participants: Physicians who participated in the intervention.
- CHV Workshop Participants: CHVs who participated in the intervention.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Physician Workshop Participants | CHV Workshop Participants | Total
Number analyzed (Participants) | 23 | 23 | 19 | 22 | 37 | 0 | 124
Age, Continuous [Mean (Full Range); unit: years] | 18.04 [15 to 23] | 18.52 [15 to 22] | 17.58 [15 to 24] | 18.91 [15 to 25] | 45.2 [26 to 67] |  | 23.65 [15 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 19 | 22 | 18 |  | 105
  Male | 0 | 0 | 0 | 0 | 19 |  | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 |  | 0
  Not Hispanic or Latino | 23 | 23 | 19 | 22 | 37 |  | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 23 | 23 | 19 | 22 | 37 |  | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 |  | 0
  White | 0 | 0 | 0 | 0 | 0 |  | 0
  More than one race | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  India | 23 | 23 | 19 | 22 | 37 |  | 87

OUTCOME MEASURES:

1. Primary Outcome: Change in Sexual and Reproductive Health and Rights Knowledge Survey Score
Description: Change from baseline to end of intervention (~10 weeks) will be measured using the subscale "Sexual and Reproductive Health Knowledge" subscale of the "Illustrative Questionnaire for Interview-Surveys with Young People" [Cleland, et al. 2001(1)], which has been validated and used to assess adolescent and young adult knowledge about sexual and reproductive health and rights. The survey consists of a subset of 22 questions, and takes approximately 20 minutes to complete. Each correct answer receives 1 point, while wrong answers and "I don't know" responses receive 0 points. The total score is the sum of responses and ranges from 0-22. Higher scores suggest better sexual and reproductive health and rights knowledge.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 0.45 (0.02) | 0.44 (0.03) | 0.47 (0.04) | 0.49 (0.04)

2. Secondary Outcome: Change in Clinic Service Uptake/Use: Change in Number of Requests for Contraception
Description: The change from baseline to end of intervention (~10 weeks) will be measured asking AGYW about their most recent healthcare usage (where they went for healthcare, the reason they went, and what services and referrals they requested). This outcome measures the change in the number of requests for contraception, and is measured across all participants.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Number; unit: Number of requests for contraception
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
Number of requests for contraception | -1 | 0 | -2 | 1

3. Secondary Outcome: Change in Clinic Service Uptake/Use: Change in Number of Requests for Menstrual Health Materials/Support (MHM/S)
Description: The change from baseline to end of intervention (~10 weeks) will be measured asking AGYW about their most recent healthcare usage (where they went for healthcare, the reason they went, and what services and referrals they requested). This outcome measures the change in the number of requests for menstrual health materials/support (MHM/S), and is measured across all participants.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Number; unit: Number of requests for MHM/S
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
Number of requests for MHM/S | -1 | 0 | -4 | -3

4. Secondary Outcome: Change in Clinic Service Uptake/Use: Change in Number of Requests for STI/HIV Tests
Description: The change from baseline to end of intervention (~10 weeks) will be measured asking AGYW about their most recent healthcare usage (where they went for healthcare, the reason they went, and what services and referrals they requested). This outcome measures the change in the number of requests for STI/HIV tests, and is measured across all participants.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Number; unit: Number of requests for STI/HIV tests
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
Number of requests for STI/HIV tests | -2 | 0 | -4 | 0

5. Secondary Outcome: Change in Personal and Community Safety
Description: The change from baseline to end of intervention (~10 weeks) will be measured asking AGYW about their perceptions of personal and community safety. These questions were developed and validated for use in India by Bhatla, et al. 2013 (2). This consists of 7 questions, and takes approximately 7 minutes to complete. Score range from 0 - 4, higher scores suggest greater feelings of safety.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | -0.14 (0.09) | -0.16 (0.15) | -0.43 (0.16) | -0.38 (0.18)

6. Secondary Outcome: Change in Gender Norms
Description: The change from baseline to end of intervention (~10 weeks) will be measured asking AGYW about their perceptions regarding what are acceptable behaviors for young men and women in their community. These questions were developed and validated for use in India by Achyut, et al. 2011 (3). This consists of 40 questions, and takes approximately 30 minutes to complete. Score ranges from 1-4, higher scores suggest more gender equitable norms.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 0.16 (0.03) | 0.06 (0.06) | 0.07 (0.07) | 0.15 (0.08)

7. Secondary Outcome: Change in Perceived Self-efficacy and Agency
Description: This is a sub-scale asking AGYW about their perceived self-efficacy and agency will be measured at baseline. These questions were developed and validated for use by Brault, et al. 2017 (4). This consists of 9 questions, and takes approximately 5 minutes to complete. Score ranges from 1-4, higher scores suggest greater self-efficacy.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 0.18 (0.03) | 0.51 (0.05) | 0.49 (0.06) | 0.46 (0.06)

8. Secondary Outcome: Change in Mental Health as Measured Using GAD-7
Description: The Generalized Anxiety Disorder 7-item (GAD-7) questionnaire is an assessment of symptoms of generalized anxiety disorder. Each item is rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-21; higher scores indicate greater presence of generalized anxiety disorder symptoms.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 0.38 (0.35) | -1.55 (0.62) | -1.92 (0.71) | -1.76 (0.80)

9. Secondary Outcome: Change in Mental Health as Measured Using PHQ-8
Description: The Patient Health Questionnaire depression scale (PHQ-8) is an 8-item assessment of depressive symptomology. The questionnaire is scored by adding up the values of all eight items on the scale. Each item uses a 4-point Likert-type scale, ranging from 0 ("not at all") to 3 ("nearly every day"). The total score ranges from 0 to 24 points, with higher scores indicating greater depressive symptomology.
Time Frame: Pre-Test (Baseline), Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 0.30 (0.29) | -0.85 (0.53) | -1.23 (0.62) | -0.98 (0.72)

10. Secondary Outcome: Intervention Acceptability as Rated by AGYW
Description: Measured at the end of the intervention (~10 weeks). These questions assess the acceptability of the intervention, and were developed by Hunsley 1992 (6). This consists of 6 questions, and takes approximately 5 minutes to complete. Score ranges from 1- 7, higher scores suggest higher intervention acceptability.
Time Frame: Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 6.81 (0.36) | 6.64 (0.44) | 6.84 (0.28) | 6.89 (0.23)

11. Secondary Outcome: Satisfaction With Intervention/Services as Rated by AGYW
Description: Measured at the end of the intervention (~10 weeks).These questions assess participant satisfaction with the intervention, and are described by Lewis, et al. 2015 (7). This consists of 11 questions, and takes approximately 10 minutes to complete. Score ranges from 1 to 12, higher scores suggest greater satisfaction with services
Time Frame: Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 8.58 (0.59) | 8.63 (0.90) | 8.48 (0.71) | 8.39 (0.69)

12. Secondary Outcome: Intervention Feasibility as Rated by AGYW
Description: Measured at the end of the intervention (~10 weeks).These questions assess participant perceptions of the feasibility of the intervention, and are described by Lewis, et al. 2015 (7). This consists of 4 questions, and takes approximately 2 minutes to complete. Score ranges from 1 to 5, higher scores suggest higher intervention feasibility.
Time Frame: Week 10 Post-Initiation of Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 23 | 23 | 19 | 22
score on a scale | 5 (0) | 4.78 (0.41) | 5 (0) | 4.96 (0.21)

ADVERSE EVENTS:
Time Frame: About 10 weeks.
Description: Note that adverse event data were not collected from Physician or CHV participants.
Groups:
- Group B: Participants in Group B have wait list control data collected during Intervention Period 1, and receive the intervention during Intervention Period 2. The adverse event/serious adverse event/mortality data represent data collected during the wait-list control period and intervention periods. These timepoints are combined as no adverse events/serious adverse events/mortality were observed.
- Group C: Participants in Group C have wait list control data collected during Intervention Period 2, and receive the intervention during Intervention Period 3. The adverse event/serious adverse event/mortality data represent data collected during the wait-list control period and intervention periods. These timepoints are combined as no adverse events/serious adverse events/mortality were observed.
- Group D: Participants in Group D have wait list control data collected during Intervention Period 3 and receive the intervention during Intervention Period 4. The adverse event/serious adverse event/mortality data represent data collected during the wait-list control period and intervention periods. These timepoints are combined as no adverse events/serious adverse events/mortality were observed.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT04307849/Prot_SAP_000.pdf